CLINICAL TRIAL: NCT00588159
Title: Preoperative Gabapentin for Acute and Chronic Post-thoracotomy Analgesia: A Randomized, Double-blinded, Placebo-controlled Study
Brief Title: Preoperative Gabapentin for Acute and Chronic Post-thoracotomy Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michelle Kinney (Other)
Responsible Party: Sponsor-Investigator, Michelle Kinney, Michelle A. O. Kinney, MD, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-004145
Record Dates: First submitted 2007-12-18; First posted 2008-01-08 (Estimated); Results first posted 2011-08-12 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-03

CONDITIONS: Pain
Keywords: Preoperative gabapentin; Acute pain; Post-thoracotomy pain; Epidural analgesia
MeSH Terms: conditions — Pain; Acute Pain | interventions — Gabapentin; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin preoperatively (Experimental): Preoperative gabapentin 600 mg orally within 2 hours prior to surgery.
  Interventions: Drug: Gabapentin
- Active placebo (Placebo Comparator): Diphenhydramine 12.5 mg orally 2 hours preoperatively.
  Interventions: Drug: Diphenhydramine

INTERVENTIONS:
Drug: Gabapentin — gabapentin 600 mg orally within 2 hours preoperatively, epidural infusion of 0.075% bupivacaine with 10 mcg/ml of hydromorphone at 6 ml/hour, fentanyl intravenous patient controlled analgesia at 10 mcg every 10 minutes as needed with a 200 mcg 4 hour lockout, oral acetaminophen 650 mg orally every 6 hours as needed for pain, intravenous ketorolac 15 mg every 6 hours as needed for pain.
  Other Names: Neurontin
  Arms: Gabapentin preoperatively
Drug: Diphenhydramine — Diphenhydramine 12.5 mg orally within 2 hours preoperatively, epidural infusion of 0.075% bupivacaine with 10 mcg/ml of hydromorphone at 6 ml/hour, fentanyl intravenous patient controlled analgesia at 10 mcg every 10 minutes as needed with a 200 mcg 4 hour lockout, oral acetaminophen 650 mg orally every 6 hours as needed for pain, intravenous ketorolac 15 mg every 6 hours as needed for pain.
  Other Names: Benadryl
  Arms: Active placebo

SUMMARY:
One dose of either gabapentin or placebo will be given to patients prior to thoracotomy. Patients will also receive an epidural infusion, intravenous patient-controlled analgesia with fentanyl, oral acetaminophen and intravenous ketorolac as needed to achieve optimal analgesia. Pain ratings and supplemental medication use will be recorded for 48 hours and will also be assessed at 3 months postoperatively to determine whether the patients who received gabapentin had improved analgesia and/or required less supplemental medication than the placebo group.

DETAILED DESCRIPTION:
The gabapentin dose utilized is 600 mg. The epidural infusion utilizes bupivacaine 0.075% with hydromorphone 10 mcg/cc infusing at 6 cc/hour. The settings for the fentanyl patient-controlled analgesia device start at 10 mcg every 10 minutes with a 200 mcg 4 hour maximum.

ELIGIBILITY:
Inclusion criteria:

* Age 45-75 years
* Undergoing thoracotomy (lobectomy, segmentectomy, wedge resection)

Exclusion criteria:

* Undergoing chest wall resection, gastroesophageal surgery
* Enrolled in another post-thoracotomy analgesic research protocol
* Pre-existing pain syndrome
* Current gabapentin or pregabalin therapy
* Inability to understand the study protocol
* Coagulopathy
* Current use of anticoagulants
* Allergy to medications on protocol
* Creatinine >1.3
* Moderate or severe aortic stenosis
* Severe psychological disorders
* Bacteremia, osteomyelitis, or infection at site of thoracic epidural placement
* History of previous thoracotomy
* Patient declines preoperative epidural catheter placement
* Prisoners or other institutionalized individuals
* Severe hepatic, renal or cardiovascular disorders
* Women who can become pregnant

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2007-06; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A. Kinney, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kinney MA, Mantilla CB, Carns PE, Passe MA, Brown MJ, Hooten WM, Curry TB, Long TR, Wass CT, Wilson PR, Weingarten TN, Huntoon MA, Rho RH, Mauck WD, Pulido JN, Allen MS, Cassivi SD, Deschamps C, Nichols FC, Shen KR, Wigle DA, Hoehn SL, Alexander SL, Hanson AC, Schroeder DR. Preoperative gabapentin for acute post-thoracotomy analgesia: a randomized, double-blinded, active placebo-controlled study. Pain Pract. 2012 Mar;12(3):175-83. doi: 10.1111/j.1533-2500.2011.00480.x. Epub 2011 Jun 16. PMID 21676165

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin Preoperatively: Preoperative gabapentin 600 mg p.o. within 2 hours prior to surgery.
- Active Placebo: Diphenhydramine 12.5 mg p.o. 2 hours preoperatively.
Period: Overall Study
Arm/Group | Gabapentin Preoperatively | Active Placebo
Started | 72 | 74
Completed | 57 | 63
Not Completed | 15 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin Preoperatively | Active Placebo | Total
Number analyzed (Participants) | 72 | 74 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 38 | 71
  >=65 years | 39 | 36 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (7) | 64 (7) | 64 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 38 | 70
  Male | 40 | 36 | 76
Region of Enrollment [Number; unit: participants]
  United States | 72 | 74 | 146

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Score at Rest
Description: Pain scores every 4 hours for 48 hours postoperatively, utilizing the numeric rating scale with 0 being no pain and 10 the most severe pain you can imagine.
Time Frame: 48 hours
Population: The number of participants analyzed included those who had successfully completed the protocol, by having received the study medication preoperatively, having received a functioning epidural prior to discharge from the postanesthesia care unit, and having undergone a thoracotomy. Numeric Rating Scale (NRS) ranges from 0 (no pain) to 10 (worst).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gabapentin Preoperatively | Active Placebo
Number analyzed (Participants) | 57 | 63
Units on a scale | 3.1 (1.9) | 2.9 (1.8)

2. Secondary Outcome: Opioid Consumption in First 24 Hours Postoperatively
Time Frame: 24 hours
Population: The number of participants analyzed included those who had successfully completed the protocol, by having received the study medication preoperatively, having received a functioning epidural prior to discharge from the postanesthesia care unit, and had a thoracotomy. Opioid use in mg is based on morphine equivalents (Hanks GW, Br J Cancer 2001).
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Gabapentin Preoperatively | Active Placebo
Number analyzed (Participants) | 57 | 63
mg | 111.9 (116.9) | 118.1 (94.7)

3. Secondary Outcome: Number of Participants With Pain at Thoracotomy Site 3 Months Postoperatively
Description: Patients were contacted at 3 months post-thoracotomy and asked if they had pain at the thoracotomy site. We observed the number of participants with the presence of pain at thoracotomy site at 3 months postoperatively.
Time Frame: 3 months postoperatively
Population: The number of participants analyzed included those who had successfully completed the protocol, by having received the study medication preoperatively, having received a functioning epidural prior to discharge from the postanesthesia care unit, and had a thoracotomy. Patients who rated their average pain 1 or greater were included.
Measure: Number; unit: Participants
Arm/Group | Gabapentin Preoperatively | Active Placebo
Number analyzed (Participants) | 57 | 63
Participants | 37 | 38

4. Primary Outcome: Average Pain Score With Coughing the First Morning Following Surgery
Description: Patients were asked on the first morning following surgery how they rated their pain with coughing utilizing the Numeric Rating Scale for pain, with 0 being no pain and 10 being the worst pain imaginable. The range is 0-10.
Time Frame: First morning following surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Gabapentin Preoperatively | Active Placebo
Number analyzed (Participants) | 57 | 63
Units on a scale | 5.2 (2.9) | 5.0 (2.6)

5. Primary Outcome: Average Pain Score With Coughing on Second Morning After Surgery
Description: Numeric rating scale pain score with coughing on second morning after surgery, range 0-10.
Time Frame: Second morning after surgery
Population: The number of participants analyzed included those who had successfully completed the protocol, by having received the study medication preoperatively, having received a functioning epidural prior to discharge from the postanesthesia care unit, and having undergone a thoracotomy.Numeric Rating Scale (NRS) ranges from 0 (no pain) to 10 (worst).
Measure: Mean (Standard Deviation); unit: Unites on a scale
Arm/Group | Gabapentin Preoperatively | Active Placebo
Number analyzed (Participants) | 57 | 63
Unites on a scale | 5.0 (2.2) | 5.1 (2.5)

6. Secondary Outcome: Opioid Consumption in Second 24 Hour Hour Period (Hours 24-48) Postoperatively
Description: Opioid equivalents (parenteral and/or oral) utilized by patient between hours 24-48 postoperatively
Time Frame: 48 hours postoperatively
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Gabapentin Preoperatively | Active Placebo
Number analyzed (Participants) | 57 | 63
mg | 114.4 (106.8) | 121.6 (110.3)

ADVERSE EVENTS:
Time Frame: 48 hours following entrance into the recovery room.
Arm/Group | Gabapentin Preoperatively | Active Placebo
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/63
Other Adverse Events (participants affected / at risk) | 4/57 | 4/63
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin Preoperatively (N=57) | Active Placebo (N=63)
Sedation (Nervous system disorders) | 4 (4) | 4 (4) — Sedation was graded by nursing staff every 4 hours using the Pain Management Sedation Scale (0=awake; 1=drowsy, dozes intermittently, easily arousable; 2=sedated, sleeps, but can be aroused; 3=difficult to arouse

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes